CLINICAL TRIAL: NCT00665522
Title: A Prospective Safety Surveillance Study of IONSYS (Fentanyl HCl)
Brief Title: A Prospective Safety Surveillance Study of Fentanyl Iontophoretic Transdermal System (40 Mcg)
Status: Terminated | Type: Observational
Why Stopped: Study was terminated at the request of the company due to the recall of marketed product in Europe.
Sponsor: Alza Corporation, DE, USA (Industry)
Responsible Party: Sponsor
Other Study IDs: CR013201; C-2006-001
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Pain
Keywords: Pain; Postoperative Analgesia; Patient-Controlled Opioids
MeSH Terms: conditions — Pain | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 001: fentanyl iontophoretic transdermal system (40mcg) No Placebo 40 mcg per dose maximum of 6 doses/hourtotal maximum 80 doses/24 hours
  Interventions: Drug: fentanyl iontophoretic transdermal system (40mcg) No Placebo
- 002: IV PCA with standard of care opioid analgesia per 24 hour period
  Interventions: Drug: IV PCA with standard of care opioid analgesia

INTERVENTIONS:
Drug: fentanyl iontophoretic transdermal system (40mcg) No Placebo — 40 mcg per dose, maximum of 6 doses/hour
  Groups: 001
Drug: IV PCA with standard of care opioid analgesia — total maximum 80 doses/24 hours
  Groups: 002

SUMMARY:
The purpose of the study is to document the use of fentanyl HCl 40 mcg system under routine conditions and obtain a more comprehensive understanding of the safety of the system and complications that may not be spontaneously reported.

DETAILED DESCRIPTION:
The safety of fentanyl HCl 40 mcg system has been evaluated in a number of research studies. Although this research included patients with acute moderate to severe pain after particular types of surgery, including abdominal, pelvic, and orthopedic procedures, the safety associated with use under conditions of routine post-operative clinical care may not have been completely characterized by the study database. This study will be a surveillance study on the risks associated with the usage of fentanyl HCl 40 mcg system under such conditions. Approximately 3,000 patients who have scheduled surgery and need treatment of acute moderate to severe post-operative pain and are treated with fentanyl HCl 40 mcg system in the hospital setting will be evaluated. In addition, a group of approximately 1,500 patients treated with opioid intravenous patient-controlled analgesia (IV PCA) will be matched to fentanyl HCl 40 mcg system patients with respect to (1) country (match will first be sought within the same research center, and extended to patients in the same country if no match is found), (2) pre-surgical physical condition and (3) surgery risk (high risk versus low risk). Patients at multiple research centers in multiple countries will be included. Patients with planned surgery and anticipated use of opioid pain management for post-operative care who are candidates for treatment with fentanyl HCl 40 mcg system or IV PCA opioid treatment will have the study explained and may participate after giving informed consent if they meet the study entry criteria. Enrollment in the study begins prior to their surgical procedure. Patients will receive treatment and care according to the standard practices at the study center, including: treatment choice, pain management set-up, and operation. Data collection in this observational (non-interventional) study will begin after informed consent is obtained and admission to the study center for the surgical procedure and will continue until discontinuation of fentanyl HCl 40 mcg system or IV PCA opioid treatment. Any significant changes in medical condition will be followed until they have resolved or have become medically stable. Patients will receive fentanyl iontophoretic transdermal system 40 mcg (fentanyl HCl 40 mcg delivered by patient activation over 10 minutes for a maximum of 6 doses/hour for up to 24 hrs or 80 total doses) or Intravenous Patient-Controlled Analgesia (IV PCA) opioid (medication choice, treatment regimen, and operation of the PCA pump to be consistent with standard practice at participating centers). Treatment duration to be determined by the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Planned surgery
* Planned use of fentanyl HCl 40 mcg system or IV Patient-Controlled Analgesia opioid treatment for postoperative pain

Exclusion Criteria:

- Pain resulting from emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 3,000 patients who have scheduled surgery and need treatment of acute moderate to severe post-operative pain and are treated with fentanyl HCl 40 mcg system in the hospital setting will be evaluated. In addition, a group of approximately 1,500 patients treated with opioid intravenous patient-controlled analgesia (IV PCA) will be matched to fentanyl HCl 40 mcg system patients with respect to (1) country (match will first be sought within the same research center, and extended to patients in the same country if no match is found), (2) pre-surgical physical condition and (3) surgery risk (high risk versus low risk). Patients at multiple research centers in multiple countries will be included.
Sampling Method: Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2007-12; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The purpose of the study is to document the use of fentanyl HCl 40 mcg system under routine conditions and obtain a more comprehensive understanding of the safety of the system and complications that may not be spontaneously reported. | Patients will receive treatment and care according to the standard practices at the study center, including: treatment choice, pain management set-up, and operation.

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — ALZA
Locations (26):
- Austria (8):
  - Feldkirch
  - Graz
  - Klagenfurt
  - Linz
  - Salzburg
  - Vienna
  - Wels
  - Wiener Neustadt
- Finland (2):
  - Helsinki
  - Kuopio
- Germany (15):
  - Aachen
  - Bad Dürkheim
  - Bergisch Gladbach
  - Berlin
  - Bonn
  - Cologne
  - Hamburg
  - Hanover
  - Kaiserslautern
  - Koblenz
  - München
  - Neubrandenburg
  - Sinsheim
  - Speyer
  - Wÿrzburg
- Sneek, Netherlands

REFERENCES:
- See also: A Prospective Safety Surveillance Study of IONSYS (Fentanyl HCl) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=116&filename=CR013201_CSR.pdf